CLINICAL TRIAL: NCT05338008
Title: Serum and Wound Vancomycin Levels Following Intrawound Administration in Primary Total Hip Arthroplasty
Brief Title: Intrawound Administration of Vancomycin in THA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Principal Investigator, Xiang Shuai, MD, Principal Investigator, The Affiliated Hospital of Qingdao University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AHQingdao VancoTHA
Record Dates: First submitted 2022-04-11; First posted 2022-04-20 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Hip

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intrawound Administration of Vancomycin (Experimental): After closure of the arthrotomy, 1 g of vancomycin powder suspended in 30ml of normal saline was injected directly into the joint with an 18-gauge needle. Then 20ml of normal saline was injected directly into the joint.
  Interventions: Procedure: Intrawound administration of vancomycin after closure of the arthrotomy
- Intrawound Administration of Vancomycin combined with epsilon-aminocaproic acid (EACA) (Experimental): After closure of the arthrotomy, 1 g of vancomycin powder suspended in 30ml of normal saline was injected directly into the joint with an 18-gauge needle. Then 4g (20ml) of epsilon-aminocaproic acid (EACA) was injected directly into the joint.
  Interventions: Procedure: Intrawound administration of vancomycin after closure of the arthrotomy
- Intrawound Administration of epsilon-aminocaproic acid (EACA) (No Intervention): After closure of the arthrotomy, 30ml of normal saline was injected directly into the joint with an 18-gauge needle. Then 4g (20ml) of epsilon-aminocaproic acid (EACA) was injected directly into the joint.

INTERVENTIONS:
Procedure: Intrawound administration of vancomycin after closure of the arthrotomy — After closure of the arthrotomy, 1 g of vancomycin powder suspended in 30ml of normal saline was injected directly into the joint with an 18-gauge needle.
  Arms: Intrawound Administration of Vancomycin; Intrawound Administration of Vancomycin combined with epsilon-aminocaproic acid (EACA)

SUMMARY:
The purpose of this study is to determine the intra-articular and serum levels of vancomycin over the first 24 hours postoperatively after intra-articular administration of a standard dose of vancomycin in primary total hip arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 18;
2. Total hip arthroplasty for advanced hip diseases including femoral neck fracture, developmental dysplasia of hip, and osteonecrosis of the femoral head.

Exclusion Criteria:

1. Diminished mental capacity
2. Vancomycin allergy
3. Chronic kidney disease stage III and stage IV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Intra-articular vancomycin concentration | 2 hours, 8 hours and 24 hours postoperatively
Serum vancomycin concentration | 2 hours, 8 hours and 24 hours postoperatively
Renal function | Postoperative Day 1 and Day 3
  blood urea nitrogen (BUN), creatinine (Cr), GFR
Blood loss | Postoperative Day 3

CONTACTS AND LOCATIONS:
Overall Officials: Shuai Xiang, M.D., Principal Investigator — The Affiliated Hospital of Qingdao University
Locations (1):
- The affiliated hospital of Qingdao University, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP
Time Frame: After completing the trial.